CLINICAL TRIAL: NCT06752720
Title: Intracerebral Autologous Mesenchymal Stem Cell Transplantation Therapy for Patients with Ischemic Stroke in Chronic Phase: Phase 2a Clinical Trial
Brief Title: Intracerebral Autologous Stem Cell Therapy for Chronic Stroke Patients
Acronym: RAINBOW-2a
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hokkaido University Hospital (Other)
Collaborators: RAINBOW Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R6-8
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Stroke, Ischemic; Stroke; Sequelae
Keywords: stem cell therapy; mesenchymal stem cell; ischemic stroke; chronic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Bronchiolitis Obliterans Syndrome | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stem cell transplantation (Experimental): Intracerbral transplantation of autologous mescenchymal stem cells (HUNS001-01, 4 x 10^7 MSC cells)
  Interventions: Drug: Stem cell Transplantation

INTERVENTIONS:
Drug: Stem cell Transplantation — Manufactured autologous mescenchymal stem cell (HUNS001-01) in our cell processing center will be injected into the brain, totally 4 x 10^7 cells, in 2 brain sites.

SUMMARY:
The goal of this clinical trial is to evaluate if autologous mesenchymal stem cell (HUNS001-01) transplantation therapy can provide neurological recovery in patients with chronic stage of stroke resulting in moderate to severe neurological sequelae. The main questions it aims to answer are:

Can HUNS001-01 intracerebral transplantation demonstrate improvement in the mRS of disability for 1 year after intervention? Can HUNS001-01 intracerebral transplantation can be performed without any adverse events for 1 year after intervention?

Participants will receive the below interventions.

* Screening for the eligibility to enroll the clinical trial (interview, blood test, imaging)
* Harvest of platelet concentrates (PC)
* Harvest of bone marrows (BM)
* Receive intracerebral transplantation surgery of HUNS001-01
* Post-operative rehabilitation
* Follow-up studies (until 1 year or termination of the trial)

ELIGIBILITY:
Inclusion criteria

1. Age between 20 and 70 years
2. Clinical diagnosis of ischemic stroke between 6 months and 5 years ago
3. Ischemic area in the territory of unilateral interanal cerebral artery
4. Moderate to severe neurological symptoms; mRS 3 or 4, and Brunnstrom stage Ⅲ or IV
5. Subjects with a DTI-RAINBOW (R-DTI) value of more than 70% at screening MR imaging
6. No significant neurological impairment before the stroke (Pre-stroke mRS of 0 or 1)
7. Subjects who can give informed consent by its self

Exclusion criteria

1. Subject showing severe lower extremity contracture (Maximum knee extension less than -15 degrees, Maximum ankle flexion less than 0 degree)"
2. Anaemia (Hg < 10·0 g/dL)
3. Thrombocytopaenia (platelet count < 100,000/mm3)
4. Severe heart disease (ischaemic heart disease, heart failure)
5. Severe Systemic organ failure ALT <3·0× upper limit of normal Total bilirubin < 1·5× upper limit of normal Serum creatinine < 1·5× upper limit of normal
6. History of malignancy
7. Carriers of infectious disease: syphilis, HBV, HCV, HIV-1/HIV-2, HTLV-1, parvovirus B19
8. Pregnant or lactating or expecting to become pregnant during the study
9. Known serious allergy to any agents used in the study
10. Contraindication for magnetic resonance imaging
11. History of seizure within 2 years
12. Subject's body weight less than 45 kg for male and 40kg for female "13. Participating in another clinical trial within 90 days, or planning to participate in another clinical trial in the future"

14. Any condition that in the judgement of the investigator would place the patient at undue risk

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of HUNS001-01 administration | one year
  The frequency of the improvement in mRS of disability by 1 or more from baseline

SECONDARY OUTCOMES:
Safety of HUNS001-01 administration | one year
  frequency of Adverse Event
Change in NIHSS examination | one year
  Mean improvement of NIHSS (0-42, higher score means worse outcome)
Change in FIM examination | one year
  Mean improvement of FIM (18-126, higher score means better outcome)
Change in Fugl-Myer examination | one year
  Mean improvement of Fugl-Myer (0-226, higher score means better outcome)
Change in Barthal index examination | one year
  Mean improvement of Barthal index (0-100, higher score means better outcome)
Change in FDG-PET examination | one year
  Mean improvement of FDG-PET set for ipsilateral motor cortex
Change in IMZ-SPECT examination | one year
  Mean improvement of IMZ-SPECT set for ipsilateral motor cortex

CONTACTS AND LOCATIONS:
Locations (1):
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: No